CLINICAL TRIAL: NCT00175578
Title: Differences in SELDI Produced Serum Protein Profiles of Non-small Cell Lung Cancer Patients Compared to Healthy Heavy Smoking Adults
Brief Title: Detection of Early Lung Cancer by Serum Protein Expression Profiling
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: C04-0640
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Early stage (0/I) non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Promising new technology exists to examine small proteins that are shed by cancers into the blood stream. The purpose of this study is to see if there are differences in the proteins and protein levels in blood from individuals with early stage lung cancer compared to healthy adults.

DETAILED DESCRIPTION:
A prospective longitudinal patient-based pilot study is proposed whereby surfaced enhanced laser desorption ionization time-of-flight mass spectroscopy (SELDI-TOF-MS) will be used to discover and validate serum proteomic expression profiles diagnostic of early lung cancer. A unique approach will be used to compare the serum proteomic expression profiles of patients with non-small cell lung cancer compared to healthy heavy smoking adults, as well as differences before and after anatomic pulmonary resection with curative intent. Discriminatory proteins will be selected by their differential expression before compared to after surgical removal of a tumor. The protein profile of blood obtained from the draining pulmonary vein at the time of resection will be used to identify materials potentially shed by the tumor that may serve as biomarkers in peripheral blood. The serum samples will be used to develop a training data set and then a test set for validation using a class prediction model. Candidate proteomic patterns will then serve as a basis for a larger prospective multi-centre clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Presence of early stage non-small cell lung cancer
* Elective surgical resection of lung lesion at Vancouver General Hospital (VGH)
* No preoperative chemoradiation therapy
* No previous cancer
* Ability to provide informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer and healthy heavy smoking adults.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2005-05; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Yee, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital BC Cancer Agency, Vancouver, British Columbia, Canada